CLINICAL TRIAL: NCT06244953
Title: Timely Interventions to Enable and Reach Patients With Heart Failure, and Their Caregivers With Palliative Care
Acronym: TIER-HF-PC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National Heart Centre Singapore (Other); Khoo Teck Puat Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TIER-HF-PC
Record Dates: First submitted 2024-01-17; First posted 2024-02-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: Palliative care; Patients; Caregivers; Distress thermometer (DT); Integrated Palliative Care Outcome Scale (IPOS); TIER-HF-PC
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular screening with needs-guided palliative care treatments (Experimental): The patient continues to receive clinical care from the cardiologist, as well as palliative care treatments that are based upon his/her reported distress and concerns.
  Interventions: Other: TIER-HF-PC
- Usual Care (Other): Patient is referred by cardiologist to palliative care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: TIER-HF-PC — The patient will be assigned to one of the three levels of care which is determined by the results given by Distress Thermometer (DT) and the Integrated Palliative Care Outcome Scale (IPOS).
  Arms: Regular screening with needs-guided palliative care treatments
Other: Usual Care — Patient continues on clinical care by his/her cardiologist. If the cardiologist picks up their symptoms or other concerns, he/or can be referred to a specialist palliative care physician by the cardiologist.
  Arms: Usual Care

SUMMARY:
There is evidence for the effectiveness and feasibility of the individual components of TIER-HF-PC, however there is a need to test how these individual components interact to allow the researchers to deliver TIER-HF-PC as a model of care in its totality. In the short term, this study will assess if TIER-HF-PC is beneficial for patients and caregivers.

DETAILED DESCRIPTION:
Timely Interventions to Enable and Reach patients with Heart Failure, and their caregivers with Palliative Care, or TIER-HF-PC, is a novel model of palliative care, designed to address gaps of palliative care delivery for patients with advanced heart failure, and their caregivers.

TIER-HF-PC is a service, led by a palliative care nurse, with support by a palliative care physician. This nurse will actively screen and monitor patients for problems, and then match the type and intensity of palliative care treatments to the severity of problems reported. The nurse will also facilitate processes for patients to initiate contact with health care providers should problems arise. This decreases the overall burden on palliative care services, enabling a scalable and more cost-effective model of care for a larger number of patients. The service will also utilize a proactive approach to care, increasing self-care skills and understanding of disease and treatment options. Earlier palliative care support will enable problems to be managed actively before they escalate into crises.

Overall aim: To test the effectiveness and implementation of the interacting components of TIER-HF-PC.

Specific aim 1a: To evaluate the impact of TIER-HF-PC on patients. The primary outcome is patient quality-of-life at 24 weeks, measured on the Kansas City Cardiomyopathy Questionnaire. Secondary outcomes include patient anxiety, depression, coping, spirituality, healthcare utilization, survival, and cost-effectiveness of TIER-HF-PC.

Specific aim 1b: To evaluate the impact of TIER-HF-PC on caregivers. Outcomes evaluated include caregiver quality-of-life.

- Hypothesis 1: The researchers hypothesize that TIER-HF-PC will be superior to usual care, in improving patient and caregiver quality-of-life.

Specific aim 2: To evaluate the implementation outcomes of TIER-HF-PC.

- Hypothesis 2: The researchers hypothesize that participants will be satisfied with the TIER-HF-PC service, though modifications might be needed for fine-tuning of the appropriateness and timeliness of care provision in TIER-HF-PC. They will evaluate these implementation outcomes through a validated service evaluation survey and semi-structured interviews. Fidelity to study protocols will be assessed through audits of case notes and study processes.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  1. 21 years or older and
  2. able to communicate in English or Chinese and
  3. be of stage C or D heart failure, as defined by American College of Cardiology/American Heart Association (ACC/AHA) classification system and
  4. have functional limitation of New York Heart Association (NYHA) functional status of at least 2 or more and
  5. be deemed by their cardiologist's clinical judgement to have an expected prognosis of at least 6 months survival, and
  6. have had a heart failure related hospitalization event (e.g. symptomatic decompensated heart failure) within 6 months prior to recruitment and
  7. have a phone that allows telecommunication.
* Caregivers must meet all the following inclusion criteria to be eligible for the study :

  * direct, unpaid, family caregiver of the patient;
  * self-reported by the patient to be the main person to be either:
  * responsible for up to 4 hours a day of caregiving tasks
  * and/or decision maker/spokesperson with the medical team
  * Caregiver may or may not live in the same residence as the patient.
  * Caregivers must be 21 years and above.
  * Able to communicate in English or Chinese.

Exclusion Criteria:

* Patients:

  1. have cognitive impairment (e.g., dementia)
  2. have severe, untreated, active mental illness (e.g., major depressive disorder)
  3. have ventricular assist device implant.
  4. have non-reversible hearing or visual loss or
  5. are active drug abuser or
  6. already known to a palliative care service.
* Caregivers who meet any of the exclusion criteria at baseline will be ineligible for the study:

  * have cognitive impairment (e.g., dementia) or
  * have severe, untreated, active mental illness (e.g., major depressive disorder)
  * have non-reversible hearing or visual loss.
  * are active drug abuser or
  * are a domestic helper for the patient

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient quality of life (QOL) | Baseline, 8 weeks, 16 weeks, and 24 weeks.
  Patient quality of life will be measured at baseline, and again at 8 weeks, 16 weeks, and 24 weeks using KCCQ-12.
  Descriptive statistics, and measures of effect size will be used to compare the study groups at baseline, 8 weeks, 16 weeks, and 24 weeks.
  Longitudinal data analyses will be conducted to examine intervention effects using linear mixed-effects-modelling for repeated measures at baseline, 8 through 16 and 24 weeks, constraining the baseline mean to be equal between intervention and control groups with indicators for time, group, and time by group interactions. Estimate of standard deviation of residuals from the mixed-effects model will be used to compute effect size (Cohen's d) to estimate the efficacy.
  The minimum score on KCCQ is 0 and maximum possible score is 100. A higher score indicates a better quality of life.

SECONDARY OUTCOMES:
Acceptability of TIER-HF-PC from patient and caregiver participants - through completion of the client satisfaction questionnaire (CSQ-4) | Up to 48 weeks.
  The total score of the CSQ-4 will be calculated for each participant. For the assessment of acceptability, scores from participants from both intervention and control groups will be pooled. The minimum expected score per participant is 4, and the maximum expected score per participant is 16. A higher score indicates higher satisfaction.
  The percentage of participants in TIER-HF-PC who have at least a CSQ score of 12 and above will also be calculated.
Patient anxiety and depression | Baseline, 8 weeks, 16 weeks, and 24 weeks.
  Patient anxiety will be tracked at baseline, 8 weeks, 16 weeks, and 24 weeks, using the hospital anxiety and depression scale (HADS). Descriptive statistics and measures of effect size will be used to compare the study groups at baseline, 8 weeks, 16 weeks and 24 weeks. Longitudinal data analyses will be conducted to examine intervention effects using linear mixed-effects-modelling for repeated measures at baseline, 8 through 16 and 24 weeks, constraining the baseline mean to be equal between intervention and control groups with indicators for time, group, and time by group interactions. Estimate of standard deviation of residuals from the mixed-effects model will be used to compute effect size (Cohen's d) to estimate the efficacy.
Patient Spirituality | Baseline, 8 weeks, 16 weeks, and 24 weeks.
  Patient spirituality will be tracked at baseline, 8 weeks, 16 weeks and 24 weeks, using the Functional Assessment of Chronic Illness Therapy Spiritual Well-Being Scale (FACIT-Sp-12). Descriptive statistics and measures of effect size will be used to compare the study groups at baseline, 8 weeks, 16 weeks and 24 weeks. Longitudinal data analyses will be conducted to examine intervention effects using linear mixed-effects-modelling for repeated measures at baseline, 8 through 16 and 24 weeks, constraining the baseline mean to be equal between intervention and control groups with indicators for time, group, and time by group interactions. Estimate of standard deviation of residuals from the mixed-effects model will be used to compute effect size (Cohen's d) to estimate the efficacy.
Caregiver Quality of Life | Baseline, 8 weeks, 16 weeks, and 24 weeks.
  The change in caregiver quality of life (QOL) at 8 weeks, 16 weeks, and 24 weeks as compared to baseline will be evaluated. The outcome measure used is the Singapore Caregiver Quality of Life Scale (SCQOLS-15). Descriptive statistics and measures of effect size will be used to compare the study groups at baseline, 8 weeks, 16 weeks and 24 weeks. Longitudinal data analyses will be conducted to examine intervention effects using linear mixed-effects-modelling for repeated measures at baseline, 8 through 16 and 24 weeks, constraining the baseline mean to be equal between intervention and control groups with indicators for time, group, and time by group interactions. Estimate of standard deviation of residuals from the mixed-effects model will be used to compute effect size (Cohen's d) to estimate the efficacy.
Assessment of impact of TIER-HF-PC on healthcare utilization | Up to 24 weeks.
  1. The difference in the number of community hospice referrals, number of emergency visits, number of intensive care visits between TIER-HF-PC participants and those in usual care will be summarized using descriptive statistics.
  2. The difference in average length of hospital admissions and average length of intensive care unit visits between TIER-HF_PC participants and those in usual care will also be summarized using descriptive statistics.
Healthcare cost analysis | Up to 24 weeks.
  The total cost of inpatient bills and outpatient bills including emergency visit bills for TIER-HF-PC participants and usual care participants from week 1 to week 24 will be summed up to quantify the cost differences between both groups by generalized linear model with Gamma model and robust standard error.
Survival analysis | Up to 48 weeks.
  The differences in survival between TIER-HF-PC and usual care will be analyzed using a Cox model regression, censoring at week 48 or death, whichever occurs earlier.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shirlyn Neo, MBBS, MRCP (UK), MMed, FAMS, Principal Investigator — National Cancer Centre, Singapore
Locations (4):
- Singapore (4):
  - National Heart Centre Singapore, Singapore
  - Sengkang General Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore
  - National Cancer Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Neo SH, Yu K, Lee CF, Cheung YB. Interventions to enable and reach patients with heart failure and their caregivers, with palliative care (TIER-HF-PC): a study protocol of a two-armed parallel group, open label randomised controlled trial that evaluates the effectiveness of a tiered model of palliative care in tertiary cardiac institutes in Singapore. BMJ Open. 2025 Mar 27;15(3):e100581. doi: 10.1136/bmjopen-2025-100581. PMID 40147986